CLINICAL TRIAL: NCT01287442
Title: Evaluation of Filtering Blebs Using the "Wuerzburg Bleb Classification Score" Compared to Other Clinical Findings, e.g. the Intraocular Pressure (IOP)
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: TE-WBCS-IOP
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Trabeculectomy — A scleral flap is created. The aqueous humor is so guided under the conjunctiva to lower IOP.

SUMMARY:
It is well established to assess the functionality of a filtering bleb by intraocular pressure (IOP), either as an absolute value or as a percent reduction, and by the need of additional antiglaucoma drugs. It is also possible to evaluate the appearance of a bleb by a clinical score, e.g. the "Wuerzburg bleb classification score" (WBCS). The purpose of this study was to find out whether there is a correlation between clinical findings, in particular IOP and the WBCS.

100 eyes within two years after trabeculectomy were included into the study. Using colour photographs the filtering bleb was evaluated according to the WBCS from two different examiners, both on different levels of clinical experience. WBCS = 1 indicates poor bleb appearance, WBCS = 15 indicates optimal bleb appearance. At the same time, clinical findings like intraocular pressure, best corrected visual acuity, slit lamp biomicroscopy and medical history were taken by another examiner.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria: Diagnosis of glaucoma, status post trabeculectomy

Exclusion criteria: age <18 Jahre, other optic neuropathy than glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of glaucoma, status post trabeculectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Study Completion 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Jens Funk, Prof. MD, Principal Investigator — University Hospital Zurich, Ophtalmic Clinic
Locations (1):
- University Hospital Zurich, Ophthalmic Clinic, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Furrer S, Menke MN, Funk J, Toteberg-Harms M. Evaluation of filtering blebs using the 'Wuerzburg bleb classification score' compared to clinical findings. BMC Ophthalmol. 2012 Jul 17;12:24. doi: 10.1186/1471-2415-12-24. PMID 22805056